CLINICAL TRIAL: NCT02943941
Title: Aquarius Pressure Variability Study
Brief Title: Pressure Variability Study
Acronym: APVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pressure
Record Dates: First submitted 2016-08-08; First posted 2016-10-25 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Other): All participants enrolled in a single arm to evaluate effect of variables (posture, respiration, exertion) on pulmonary artery pressure (PAP)
  Interventions: Other: Reveal LINQ ICM Cardiac Monitor, taped on the subject's chest rather than inserted in the body.

INTERVENTIONS:
Other: Reveal LINQ ICM Cardiac Monitor, taped on the subject's chest rather than inserted in the body. — Cardiac Monitor with LINQ™ HF Investigational RAMware download
  Other Names: Interventions included: Changing posture, changing respiration, and changing exertion

SUMMARY:
The purpose of this study is to understand how the pressure in the pulmonary artery changes under different conditions of posture, respiration and exertion.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study with enrollment up to 30 subjects at 2 U.S. sites. All study data can be collected on a single day as a one-time visit (lasting approximately 90-120 minutes).

This study is a Non-Significant Risk (NSR) Investigational Device Exemption (IDE) study as LINQ™ HF investigational RAMware is required to activate additional sensors in the Reveal LINQ ICM.

The patient will come to the clinic for a single in-office visit. PA pressure will be measured while the patient is in a variety of positions and during different respiratory exercises and after brief exertion. Data will be collected on eCRFs.

The effects of the different postures, respiration and exertion will be quantified using descriptive statistics (mean, standard deviation).

ELIGIBILITY:
Inclusion Criteria:

* Investigator believes the patient's condition is sufficiently stable to safely participate in the study procedures
* Subject is currently implanted with a commercially available pulmonary artery pressure sensor and device communication has been reliable (recent history of successful communications with patient communication system)

Exclusion Criteria:

* Subject has a history of primary PAH

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Verla Laager, Study Director — Medtronic
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - The Lindner Research Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Design: Single arm (all participants)
Period: Overall Study
Arm/Group | Single Arm Design
Started (All participants) | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Single arm
Arm/Group | Single Arm
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Pulmonary Artery Pressure (PAP) Due to Change in Posture
Description: Posture defined as lying left side down compared to baseline supine
Time Frame: Same day as enrollment (during office visit, maximum of 30 minutes after baseline masurement)
Population: Only 14 patients able to provide data to contribute to analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Single Arm Design: Single arm
Arm/Group | Single Arm Design
Number analyzed (Participants) | 14
mmHg | 27.7 (10.3)
Statistical Analysis 1: Comparison: Single Arm Design; Test type: Other; p = 0.429, ANOVA

2. Secondary Outcome: Change in PAP During Change in Respiration
Description: Outcome measure defined as PAP during coughing compared to PAP during normal breathing respiration at baseline.
Time Frame: Same day as enrollment (during office visit, maximum of 30 minutes after baseline measurement)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Arm
Number analyzed (Participants) | 16
mmHg | 25.9 (13.3)
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.059, ANOVA — Pressure during coughing versus normal breathing initially measured at baseline

3. Secondary Outcome: Change in PAP as Measured After Mild Exertion Compared to Initial Baseline PAP at Rest.
Time Frame: Same day as enrollment (during office visit, maximum of 10 minutes after baseline measurement)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Single Arm Design
Number analyzed (Participants) | 14
mmHg | 27.7 (12.2)
Statistical Analysis 1: Comparison: Single Arm Design; Test type: Other; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes